CLINICAL TRIAL: NCT01107015
Title: Mobile Diabetes Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HP-00041426
Record Dates: First submitted 2010-04-17; First posted 2010-04-20 (Estimated); Results first posted 2018-03-01 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2019-12

CONDITIONS: Diabetes
Keywords: Diabetes; Glucose control; Diabetes monitoring; Care management; Electronic communication; Mobile phone technology; Self care
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1: Usual Care (No Intervention): Provider-driven care, based in office, no special diabetes management; Patient self-monitoring of blood glucose (SMBG)
- Group 2: patient intervention (Active Comparator): Home diabetes monitoring by patient using mobile phone to communicate information and receive feedback
  Interventions: Device: Tailored Patient Intervention
- Group 3: patient-physician intervention (Active Comparator): Home diabetes monitoring by patient using mobile phone to communicate and receive feedback; Physician can access unanalyzed information from the patient's electronic logbook
  Interventions: Device: Patient-physician intervention
- Group 4: data analyzed intervention (Active Comparator): Home diabetes monitoring by patient using mobile phone to communicate information and receive feedback; Physician can access raw and analyzed patient data; Physician receives report summary and treatment recommendations
  Interventions: Device: Patient and PCP intervention with analyzed data

INTERVENTIONS:
Device: Tailored Patient Intervention — Patients select one of two mobile phone models, receive a one-year unlimited mobile phone data and phone service plan, receive the study treatment phone software and have access to the web-based individual patient portal. Given system-driven guidance on when to test blood glucose (bg) based on disease status, medication regimen, and time of poorest control. Patients enter bg data, carbohydrates consumed, diabetes medications taken and miscellaneous comments regarding diabetes self-care. Messages are sent to the patient's mobile phone giving feedback on entered data. Entered data are captured in real-time in the web-based logbook. Patients may provide their PCPs with printed copies of their logbooks and other information but physicians do not have access to the patient portal system. Patient action plans summarizing the patient-entered data and identifying possible self-management actions for improving their diabetes control are electronically sent to the patients every 2.5 months.
  Arms: Group 2: patient intervention
Device: Patient-physician intervention — Patients select one of two mobile phone models, receive a one-year unlimited mobile phone data and phone service plan, receive the study treatment phone software and have access to the web-based individual patient portal. Given system-driven guidance on when to test blood glucose (bg) based on disease status, medication regimen, and time of poorest control. Patients enter bg data, carbohydrates consumed, diabetes medications taken and miscellaneous comments regarding diabetes self-care. Messages are sent to the patient's mobile phone giving feedback on entered data. Entered data are captured in real-time in the web-based logbook. PCPs are provided access to a web portal where they may choose to review their patients' electronic logbooks. This is "raw" patient data that have not been analyzed.
  Arms: Group 3: patient-physician intervention
Device: Patient and PCP intervention with analyzed data — Patients select one of two mobile phone models, receive a one-year unlimited mobile phone data and phone service plan, receive the study treatment phone software and have access to the web-based individual patient portal. Given system-driven guidance on when to test blood glucose (bg) based on disease status, medication regimen, and time of poorest control. Patients enter bg data, carbohydrates consumed, diabetes medications taken and miscellaneous comments regarding diabetes self-care. Messages are sent to the patient's mobile phone giving feedback on entered data. Entered data are captured in real-time in the web-based logbook. PCPs are provided access to a secure web portal where they can see their patients' electronic logbooks. PCPs are provided with data analysis reports. The PCP is reminded that all data analysis is based on patient-entered, unvalidated data. The PCP has the option to use this information and remains responsible for all treatment decisions.
  Arms: Group 4: data analyzed intervention

SUMMARY:
The Mobile Diabetes Intervention Study trial is evaluating a diabetes coaching system, using mobile phones and patient/ physician internet portals to allow patient-specific treatment and communication by their primary care physician. We hypothesize that timely information provided to patients and their physicians can result in reduction of A1c over 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic [patient]
* A1c equal to or greater than 7.5 [patient]
* 18-64 years of age at time of recruitment [patient]
* Access to the internet (does not need to be at their home, elsewhere is fine e.g. work) [patient]
* E-mail account [patient]
* Must speak English [patient]

Exclusion Criteria:

* No insulin pump [patient]
* No current alcohol or drug abuse- must be sober 1 year [patient]
* Not currently pregnant [patient]
* No terminal diagnosis [patient]
* No dementia or Alzheimer's [patient]
* No active chemotherapy [patient]
* No significant hearing impairment [patient]
* Poorly corrected vision that would impede use of phone [patient]
* No mute or aphasia [patient]
* No diagnosis of schizophrenia, bipolar disorder, or major psychosis [patient]
* No Medicaid or Medicare
* No uninsured

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 213 (Actual)
Dates: Start 2008-06; Primary Completion 2010-08 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geppi, Study Director — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States

REFERENCES:
- [Background] Quinn CC, Gruber-Baldini AL, Shardell M, Weed K, Clough SS, Peeples M, Terrin M, Bronich-Hall L, Barr E, Lender D. Mobile diabetes intervention study: testing a personalized treatment/behavioral communication intervention for blood glucose control. Contemp Clin Trials. 2009 Jul;30(4):334-46. doi: 10.1016/j.cct.2009.02.004. Epub 2009 Feb 27. PMID 19250979
- [Derived] Quinn CC, Swasey KK, Torain JM, Shardell MD, Terrin ML, Barr EA, Gruber-Baldini AL. An mHealth Diabetes Intervention for Glucose Control: Health Care Utilization Analysis. JMIR Mhealth Uhealth. 2018 Oct 15;6(10):e10776. doi: 10.2196/10776. PMID 30322839
- [Derived] Quinn CC, Butler EC, Swasey KK, Shardell MD, Terrin MD, Barr EA, Gruber-Baldini AL. Mobile Diabetes Intervention Study of Patient Engagement and Impact on Blood Glucose: Mixed Methods Analysis. JMIR Mhealth Uhealth. 2018 Feb 2;6(2):e31. doi: 10.2196/mhealth.9265. PMID 29396389
- [Derived] Quinn CC, Swasey KK, Crabbe JCF, Shardell MD, Terrin ML, Barr EA, Gruber-Baldini AL. The Impact of a Mobile Diabetes Health Intervention on Diabetes Distress and Depression Among Adults: Secondary Analysis of a Cluster Randomized Controlled Trial. JMIR Mhealth Uhealth. 2017 Dec 7;5(12):e183. doi: 10.2196/mhealth.8910. PMID 29217502
- See also: Quinn CC, Shardell MD, Terrin ML, Barr EA, Ballew SH, Gruber-Baldini AL. Cluster-randomized trial of a mobile phone personalized behavioral intervention for blood glucose control.Diabetes Care. 2011 Sep;34(9):1934-42. Epub 2011 Jul 25. — http://www.ncbi.nlm.nih.gov/pubmed/21788632

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 2: Patient Intervention: Home diabetes monitoring by patient using mobile phone to communicate information and receive feedback
  Patients may provide their PCPs with printed copies of their logbooks and other information but physicians do not have access to the patient portal system. Patient action plans summarizing the patient-entered data and identif
- Group 3: Patient-physician Intervention: Home diabetes monitoring by patient using mobile phone to communicate and receive feedback; Physician can access unanalyzed information from the patient's electronic logbook
  PCPs are provided access to a web portal where they may choose to review their patients' electronic logbooks. This is "raw" patient data that have not be
- Group 4: Data Analyzed Intervention: Home diabetes monitoring by patient using mobile phone to communicate information and receive feedback; Physician can access raw and analyzed patient data; Physician receives report summary and treatment recommendations
  Patient and PCP intervention with analyzed data: Messages are sent to the patient's mobile phone giving feedback on entered data. Entered data are captured in real-time in the web-based logbook. PCPs are provided access to a secure web portal where they can see their patients' electro
Period: Overall Study
Arm/Group | Group 1: Usual Care | Group 2: Patient Intervention | Group 3: Patient-physician Intervention | Group 4: Data Analyzed Intervention
Started | 62 | 38 | 33 | 80
Completed | 56 | 23 | 22 | 62
Not Completed | 6 | 15 | 11 | 18

BASELINE CHARACTERISTICS:
Groups:
- Group 2: Patient Intervention: Home diabetes monitoring by patient using mobile phone to communicate information and receive feedback
  Tailored Patient Intervention: Patients enter bg data, carbohydrates consumed, diabetes medications taken. Messages are sent to the patient's mobile phone giving feedback on entered data. Entered data are captured in real-time in the web-based logbook. Patients may provide their PCPs with printed copies of their logbooks and other information but physicians do not have access to the patient portal system. Patient action plans summarizing the patient-entered data and identifying possible self-management actions for improving their diabetes control are electronically sent to the patients every 2.5 months.
- Group 3: Patient-physician Intervention: Home diabetes monitoring by patient using mobile phone to communicate and receive feedback; Physician can access unanalyzed information from the patient's electronic logbook
  Patient-physician intervention: . Patients enter bg data, carbohydrates consumed, diabetes medications taken and miscellaneous comments regarding diabetes self-care. Messages are sent to the patient's mobile phone giving feedback on entered data. PCPs are provided access to a web portal. This is "raw" patient data that have not been analyzed.
- Group 4: Data Analyzed Intervention: Home diabetes monitoring by patient using mobile phone to communicate information and receive feedback; Physician can access raw and analyzed patient data; Physician receives report summary and treatment recommendations
  Patient and PCP intervention with analyzed data:Patients enter bg data, carbohydrates consumed, diabetes medications taken and miscellaneous comments regarding diabetes self-care. Messages are sent to the patient's mobile phone giving feedback on entered data. Entered data are captured in real-time in the web-based logbook. PCPs are provided access to a secure web portal where they can see their patients' electro
- Total: Total of all reporting groups
Arm/Group | Group 1: Usual Care | Group 2: Patient Intervention | Group 3: Patient-physician Intervention | Group 4: Data Analyzed Intervention | Total
Number analyzed (Participants) | 56 | 23 | 22 | 62 | 163
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 56 | 23 | 22 | 62 | 163
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (8.4) | 52.8 (8.0) | 53.7 (8.2) | 52.0 (8.0) | 52.8 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 11 | 10 | 31 | 80
  Male | 28 | 12 | 12 | 31 | 83
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 27 | 10 | 10 | 17 | 64
  White | 26 | 12 | 9 | 39 | 86
  More than one race | 3 | 1 | 3 | 6 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 56 | 23 | 22 | 62 | 163
HbA1c [Mean (Standard Deviation); unit: percentage of HbA1c] | 9.2 (1.7) | 9.3 (1.8) | 9.0 (1.8) | 9.9 (2.1) | 9.4 (2.0)

OUTCOME MEASURES:

1. Primary Outcome: HBA1c at One Year
Time Frame: one year
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Groups:
- Group 2: Patient Intervention: Home diabetes monitoring by patient using mobile phone to communicate information and receive feedback
  Tailored Patient Intervention: Patients enter bg data, carbohydrates consumed, diabetes medications taken and miscellaneous comments regarding diabetes self-care. Messages are sent to the patient's mobile phone giving feedback on entered data. Entered data are captured in real-time in the web-based logbook. Patients may provide their PCPs with printed copies of their logbooks and other information but physicians do not have access to the patient portal system. Patient action plans summarizing the patient-entered data and identifying possible self-management actions for improving their diabetes control are electronically sent to the patients every 2.5 months.
- Group 3: Patient-physician Intervention: Home diabetes monitoring by patient using mobile phone to communicate and receive feedback; Physician can access unanalyzed information from the patient's electronic logbook
  Patient-physician intervention: Patients enter bg data, carbohydrates consumed, diabetes medications taken and miscellaneous comments regarding diabetes self-care. Messages are sent to the patient's mobile phone giving feedback on entered data. Entered data are captured in real-time in the web-based logbook. PCPs are provided access to a web portal where they may choose to review their patients' electronic logbooks. This is "raw" patient data that have not been analyzed.
- Group 4: Data Analyzed Intervention: Home diabetes monitoring by patient using mobile phone to communicate information and receive feedback; Physician can access raw and analyzed patient data; Physician receives report summary and treatment recommendations
  Patient and PCP intervention with analyzed data: Patients enter bg data, carbohydrates consumed, diabetes medications taken and miscellaneous comments regarding diabetes self-care. Messages are sent to the patient's mobile phone giving feedback on entered data. Entered data are captured in real-time in the web-based logbook. PCPs are provided access to a secure web portal where they can see their patients' electronic logbooks. PCPs are provided with data analysis reports. The PCP is reminded that all data analysis is based on patient-entered, unvalidated data. The PCP has the option to use this information and remains responsible for all treatment decisions.
Arm/Group | Group 1: Usual Care | Group 2: Patient Intervention | Group 3: Patient-physician Intervention | Group 4: Data Analyzed Intervention
Number analyzed (Participants) | 56 | 23 | 22 | 62
percentage of HbA1c | 8.5 (1.8) | 7.7 (1.0) | 7.9 (1.4) | 7.9 (1.7)
Statistical Analysis 1: Comparison: Group 1: Usual Care vs Group 2: Patient Intervention vs Group 3: Patient-physician Intervention vs Group 4: Data Analyzed Intervention; Linear mixed-effects models were used to compare mean changes in primary and secondary outcomes between UC and each active intervention. The primary analysis examined 12-month changes for glycated hemoglobin. Secondary analyses jointly compared 3-, 6-, 9-, and 12-month changes between groups. Random effects accounted for within-practice clustering and within-patient correlation; Test type: Other — Sample size was determined on the basis of the primary outcome, change in glycated hemoglobin. The comparison of UC, which included 56 patients from nine practices, to CPDS, which included 62 patients from seven practices, had 80% power to detect a difference in mean glycated hemoglobin changes of 0.65 SD, corresponding to 1.0% if SD was 1.58%, using a two-sided test with 0.05 type I error after accounting for a within cluster correlation of 0.10; p = 0.027, Mixed Models Analysis — CO (P = 0.027) and CPP (0.40) mean HbA1c levels decreased over 12 months
Statistical Analysis 2: Comparison: Group 1: Usual Care vs Group 4: Data Analyzed Intervention; Linear mixed-effects models were used to compare mean changes in primary and secondary outcomes between UC and each active intervention. The primary analysis examined 12-month changes for glycated hemoglobin; Test type: Superiority; p = 0.001, Mixed Models Analysis; Mean Difference (Net) = 0.05

ADVERSE EVENTS:
Time Frame: One year intervention period.
Description: Participants were contacted monthly to inquire about adverse events.
Arm/Group | Group 1: Usual Care | Group 2: Patient Intervention | Group 3: Patient-physician Intervention | Group 4: Data Analyzed Intervention
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/38 | 0/33 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/38 | 0/33 | 0/80
Other Adverse Events (participants affected / at risk) | 0/62 | 0/38 | 0/33 | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No